CLINICAL TRIAL: NCT06460194
Title: Botulinum Toxin A in the Treatment of Frostbite Sequelae - a Randomized, Double Blind, Placebo-controlled Study
Brief Title: Treatment of Frostbite Sequelae With Botulinum Toxin A
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No Participants Enrolled.
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018/1961(REK)
Record Dates: First submitted 2019-03-14; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Cold Hypersensitivity; Vascular System Injuries; Vibration; Disorder; Sensory Disorders; Pain, Nerve
Keywords: cold hypersensitivity; cold intolerance; vasospastic disorder; Raynauds phenomenon; botulinum toxin; infrared thermography; Quantative sensory testing
MeSH Terms: conditions — Cold Hypersensitivity; Vascular System Injuries; Sensation Disorders; Neuralgia; Raynaud Disease | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: The methodology uses a two armed, randomized, double-blind, placebo-controlled studydesign, . All participating soldiers will get two injections, one first injection at inclusion and a second injection after 6 weeks. The injections contain either BTX
  -A or an inert placebo. Both patient and treating doctor is blinded to content of the injection.
  The two patients in the primary treatment group will receive Botox at their first injection at inclusion, while the two patients in the secondary group will receive placebo as their first injection at inclusion. At 6 weeks follow up, the patients in the primary treatment group will receive their second injection of botox. The patients in the secondary treatment group now will receive their second injection, but this will be their first injection of Botox, given at their 6 weeks follow-up.
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botulinum toxin (Active Comparator): 100 IU botulinum toxin injection in the palm of the hand
  Interventions: Drug: Botuinum toxin
- Placebo (Placebo Comparator): Saline injection in the palm of the hand
  Interventions: Drug: Botuinum toxin

INTERVENTIONS:
Drug: Botuinum toxin — Injection of botulinum toxin in the palm of the hand
  Other Names: Botox

SUMMARY:
Background Digital vasospasm as part of frostbite sequelae is comparable to the vasospastic disorders found in Raynaud's phenomenon which has been successfully treated with Botulinum toxin type A injections in the palm of the hands.

Aim of this pilot study To investigate the effect of Botulinum toxin type A for frostbite sequelae in the fingers.

Hypothesis The null hypothesis which is that all study-subjects will have equal distribution of symptoms and measurements after treatment, regardless of injection with Botulinum toxin type A or placebo.

Methodology A randomized, double-blind, placebo-controlled study design, The study population consists of four patients with frostbite sequelae. The patients are randomized to either treatment with Botulinum toxin type A or placebo Two patients in the primary treatment group will receive Botulinum toxin type A at their first injection at inclusion, while the two patients in the secondary treatment group will receive normal saline (placebo) as their first injection at inclusion. At 6 weeks follow up, the primary treatment group will receive their second injection of Botulinum toxin type A and the secondary treatment group now will receive their second injection, but this will be their first injection of Botulinum toxin type A.

By using the described study-design, all participating soldiers will get treatment. However, the secondary treatment group will have a delayed onset of treatment with Botulinum toxin type A and serves as a control for the primary treatment group during the initial 6 weeks observation.

Botulinum toxin A and placed will be injected near the neurovascular bundle at the A1 pulley in the palm of the hand using a total dosage 100 U per hand (concentration 50 U per ml), 8-12 U/ injection site.

The effect of Botulinum toxin type A on subjective symptoms will be measured by Patients Subjective Symptom Score (PSSS) The effect of Botulinum toxin type A on peripheral microcirculation will be evaluated with dynamic infrared thermography (DIRT) of the dorsal side of the hands. Quantitative sensory testing will be used to evaluate the effect of Botulinum toxin type A on peripheral nerve function. Both DIRT and QST will be performed prior to the treatment with Botulinum toxin type A and placebo at the start of the pilot study, at 6 weeks as well as 6 weeks after the last injections.

Statistical methods and data analysis will be performed according to the EMA guidelines for biostatistics. Statistical analysis will be performed according to the null hypothesis.

DETAILED DESCRIPTION:
Background Frostbite sequelae can have a significant negative impact on quality of life. Depending on the type of frostbite, sequelae such as cold hypersensitivity, sensory loss, chronic pain, hyperhidrosis, growth plate disturbances and osteoarthritis may develop. Long-term paraesthesia with occasional electric shock-type sensations have also been repored. The pathophysiology of these sequelae is still poorly understood although peripheral neurovascular dysfunction plays an important role. This may result in a vasospastic disorder similar as in Raynaud's phenomenon.

Recently, the use of Botulinum toxin type A (BTX-A) for the treatment of vasospastic disorders of the hand has shown to result in great benefits for the patients by reducing the severity and number of vasospastic disorders. BTX-A injections are targeting the neurovascular bundle at or slightly proximal to the A1 pulley in the palm of the hand.

A case history has described the off-label use of BTX-A to treat a Norwegian soldier who suffered from long-term sequelae of frostbite to his hands after a military exercise. He was successfully treated with BTX-A injections in each palm of the hand. At follow up, the patient reported less pain, warmer hands and improved sensory function. Dynamic Infrared thermography (DIRT) showed improved rewarming of all fingers compared to the pre-treatment examination, while Quantattive sensory testing (QST) showed a normalization of sensory function.

Aim of this pilot study To investigate the effect of Botulinum toxin type A for frostbite sequelae in fingers.

Hypothesis The null hypothesis is that all study-subjects will have equal distribution of symptoms and measurements after treatment, regardless of injection with Botulinum toxin type A or placebo.

Methodology A two armed, randomized, double-blind, placebo-controlled study design, performed at one single centre will be used. The study population consists of four soldiers with frostbite sequelae who will be recruited from the Norwegian Armed Forces Health Registry. These four soldiers are randomized to either treatment with Botulinum toxin type A or placebo according to computer-generated random numbers provided by the research unit at the University Hospital of North Norway. Two soldiers in the primary treatment group will receive Botulinum toxin type A at their first injection at inclusion, while the two soldires in the secondary treatment group will receive normal saline (placebo) as their first injection at inclusion. At 6 weeks follow up, the primary treatment group will receive their second injection of Botulinum toxin type A and the secondary treatment group now will receive their second injection, but this will be their first injection of Botulinum toxin type A.

By using the described study-design, all participating soldiers will get treatment. However, the secondary treatment group will have a delayed onset of treatment with Botulinum toxin type A and serves as a control for the primary treatment group during the initial 6 weeks observation.

Botulinum toxin A and placed will be injected near the neurovascular bundle at the A1 pulley in the palm of the hand using a total dosage 100 U per hand (concentration 50 U per ml), 8-12 U/ injection site.

The effect of BTX- A on peripheral microcirculation will be evaluated with dynamic infrared thermography (DIRT) of the dorsal side of the hands. DIRT of the dorsal side of the hands encompass a pre-cooling phase (T1), a cooling phase of one minute (T2), and a four-minute recovery phase (T3, T4, T5 and T6). The pre-cooling phase include baseline measurements before the DIRT takes place and includes also the time from the initial image (T1) until the hands are immersed in water.

The DIRT procedure follows international standards and recommendations involving a cold challenge followed by a rewarming phase with both hands were positioned palms down on a grid made of thin nylon netting strung on a plastic frame. The nylon grid is positioned 7 cm (+/- 0.5 cm) above a uniformly heated base plate (40 +/-2°C) to ensure a thermally uniform background for the thermal imaging.

Quantitative sensory testing will be used to evaluate the effect of BTX- A on peripheral nerve function. Thermal tests will be performed with a device TSA (Medoc, Israel) attaching a thermode to the investigated body part. Thermal tests include detection thresholds for warm and cold sensation, sensory limen (i.e., perception of changing temperatures, pain thresholds for heat and cold pain as well paradoxical cold or heat sensation. It is important to notice, that the maximum temperatures produced by the device are 0° or 50° for cold and warm, respectively. The test system automatically cancels the run, when the participant did not respond with pain up to these temperatures. Mechanical tests include also detection thresholds and pain thresholds. Mechanical detection is evaluated by von Frey hairs (pressure) and a standardized tuning fork (vibration). Pain thresholds are assessed by pin prick stimulation, pressure algometry. Additional tests for allodynia are included as well. Finally, there is a test to assess temporary summation using wind-up ratio to a repeated stimulation with pinprick (10 stimuli with 1/s).

Both DIRT and QST will be performed prior to the treatment with BTX- A and placebo at the start of the pilot study, at 6 weeks as well as 6 weeks after the last injections. At 6 months follow up after the first injection DIRT and QST will be repeated again.

The patient's subjective symptoms are monitored by comparing Patient-Subjective-Symptom-Score (PSSS) after 6 weeks with the baseline values for each patient.

Statistical methods and data analysis will be performed according to the EMA guidelines for biostatistics. Statistical analysis will be performed according to the null hypothesis.

ELIGIBILITY:
Inclusion Criteria:- Sequela following 2nd degree frostbite injury in the Norwegian Armed Forces

* Entering the Norwegian Armed Forces Health Registry (NAFHR) between 01.01.2010-31.12.2014
* Still suffering from sequelae related to frostbite injury in their fingers at least four years after their initial frostbite
* Have agreed on receiving a request to participate in the NAFHR quality assurance study.

Exclusion Criteria:- Patients who do not return the signed informed consent form

* Patients who cannot read Norwegian information or answer questions in the study
* Patients who are unable to comply the examination and treatment procedures
* Patients who are unable to travel to University Hospital North Norway in Tromsø for examination and treatment
* Patients who have undergone/is undergoing surgical treatment of hands/fingers
* Patients with known allergy/anaphylaxis in relation to the injection of BTX-A
* Patients who have used/are using drugs that interact with BTX-A injection (anticoagulants)
* Patients who are pregnant before start of the trial and/or during the trial

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Subjective symptoms between injection of Botox and placebo at 6 weeks follow up | 6 weeks
  According to clinical experience, the patient s experience improvement in subjective symptoms after 4-6 weeks follow-up. The patient's subjective symptoms are monitored in a questionnaire of neurological and vasoactive sensations by comparing Patient-Subjective-Symptom-Score (PSSS) wustionnaire after 6 weeks with the baseline values for each patient.
Rewarming before and 6 weeks after treatment with Botulinum toxin | 6 weeks
  According to clinical experience, an improvement is found in the rewarming ability after 4-6 weeks follow-up after injection of Botox. The patients rewarming ability is monitored by comparing the results from Dynamic Infrared Thermography (DIRT) after 6 weeks with the baseline values for each patient.
  The DIRT examines the dynamic regulation of peripheral micro-vascularization. Examination of the dorsal side of the hands encompasses a pre-cooling phase (T1), a cooling phase with hands immersed in water for one minute (T2), and a four-minute recovery phase (T3, T4, T5 and T6).

CONTACTS AND LOCATIONS:
Overall Officials: Arne J Norheim, PhD, Principal Investigator — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schaefer G, Huguet J, Zhu SY, Plassmann P, Ring F. Adopting the DICOM standard for medical infrared images. Conf Proc IEEE Eng Med Biol Soc. 2006;2006:236-9. doi: 10.1109/IEMBS.2006.259523. PMID 17946389
- [Result] Iorio ML, Masden DL, Higgins JP. Botulinum toxin A treatment of Raynaud's phenomenon: a review. Semin Arthritis Rheum. 2012 Feb;41(4):599-603. doi: 10.1016/j.semarthrit.2011.07.006. Epub 2011 Aug 24. PMID 21868066
- [Result] Imray C, Grieve A, Dhillon S; Caudwell Xtreme Everest Research Group. Cold damage to the extremities: frostbite and non-freezing cold injuries. Postgrad Med J. 2009 Sep;85(1007):481-8. doi: 10.1136/pgmj.2008.068635. PMID 19734516
- [Result] Fabregat G, De Andres J, Villanueva-Perez VL, Asensio-Samper JM. Subcutaneous and perineural botulinum toxin type a for neuropathic pain: a descriptive review. Clin J Pain. 2013 Nov;29(11):1006-12. doi: 10.1097/AJP.0b013e31827eafff. PMID 23370086
- [Result] Norheim AJ, Mercer J, Musial F, de Weerd L. A new treatment for frostbite sequelae; Botulinum toxin. Int J Circumpolar Health. 2017;76(1):1273677. doi: 10.1080/22423982.2016.1273677. PMID 28452678
- [Result] Segreto F, Marangi GF, Cerbone V, Persichetti P. The Role of Botulinum Toxin A in the Treatment of Raynaud Phenomenon. Ann Plast Surg. 2016 Sep;77(3):318-23. doi: 10.1097/SAP.0000000000000715. PMID 26808752
- [Result] Arnold PB, Campbell CA, Rodeheaver G, Merritt W, Morgan RF, Drake DB. Modification of blood vessel diameter following perivascular application of botulinum toxin-A. Hand (N Y). 2009 Sep;4(3):302-7. doi: 10.1007/s11552-009-9169-8. Epub 2009 Feb 5. PMID 19194764
- [Result] Ring EF, Ammer K. Infrared thermal imaging in medicine. Physiol Meas. 2012 Mar;33(3):R33-46. doi: 10.1088/0967-3334/33/3/R33. Epub 2012 Feb 28. PMID 22370242
- [Result] Moreira DG, Costello JT, Brito CJ, Adamczyk JG, Ammer K, Bach AJE, Costa CMA, Eglin C, Fernandes AA, Fernandez-Cuevas I, Ferreira JJA, Formenti D, Fournet D, Havenith G, Howell K, Jung A, Kenny GP, Kolosovas-Machuca ES, Maley MJ, Merla A, Pascoe DD, Priego Quesada JI, Schwartz RG, Seixas ARD, Selfe J, Vainer BG, Sillero-Quintana M. Thermographic imaging in sports and exercise medicine: A Delphi study and consensus statement on the measurement of human skin temperature. J Therm Biol. 2017 Oct;69:155-162. doi: 10.1016/j.jtherbio.2017.07.006. Epub 2017 Jul 18. PMID 29037377
- [Result] Maier C, Baron R, Tolle TR, Binder A, Birbaumer N, Birklein F, Gierthmuhlen J, Flor H, Geber C, Huge V, Krumova EK, Landwehrmeyer GB, Magerl W, Maihofner C, Richter H, Rolke R, Scherens A, Schwarz A, Sommer C, Tronnier V, Uceyler N, Valet M, Wasner G, Treede DR. Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): somatosensory abnormalities in 1236 patients with different neuropathic pain syndromes. Pain. 2010 Sep;150(3):439-450. doi: 10.1016/j.pain.2010.05.002. PMID 20627413
- [Result] Aru RG, Songcharoen SJ, Seals SR, Arnold PB, Hester RL. Microcirculatory Effects of Botulinum Toxin A in the Rat: Acute and Chronic Vasodilation. Ann Plast Surg. 2017 Jul;79(1):82-85. doi: 10.1097/SAP.0000000000001054. PMID 28509693